CLINICAL TRIAL: NCT03738839
Title: A Comparative Assessment of Orthodontic Treatment Outcomes Using the Quantitative Light-Induced Fluorescence (QLF) Method Between Direct Bonding and Indirect Bonding Techniques in Adolescents
Brief Title: A Comparative Assessment of Orthodontic Treatment Outcomes Using the Quantitative Light-Induced Fluorescence Method
Acronym: QLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ahmet Yağcı, Ass. Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: TSA-11-3585
Record Dates: First submitted 2018-10-24; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: White Spot Lesion of Tooth; Orthodontic Malocclusion
Keywords: White Spot Lesions; Direct Bonding; Indirect Bonding; Quantitative Light-Induced Fluorescence
MeSH Terms: interventions — Quantitative Light-Induced Fluorescence; Sondhi Indirect Bonding Resin

STUDY DESIGN:
Intervention Model Description: Random sequence generation was performed with a computerized random 1:1 allocation using block sizes of 4.
Who Masked: Participant, Outcomes Assessor
Masking Description: It was not possible for the clinicians and their interventions to be blocked. The patients and the specialists were blinded to the treatment groups when their treatment groups were aware.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct Bonding (Experimental): On the individual teeth Conventional bracket placement Use conventional composite
  Interventions: Device: Quantitative Light-Induced Fluorescence; Procedure: Direct bonding
- Indirect bonding (Experimental): On the dental stone models Indirect bracket placement Use flowable composite Use transfer trays
  Interventions: Device: Quantitative Light-Induced Fluorescence; Procedure: Indirect bonding
- Quantitative Light-Induced Fluorescence (Active Comparator): Use special device and software Determination of the number and effect of caries
  Interventions: Device: Quantitative Light-Induced Fluorescence; Procedure: Direct bonding; Procedure: Indirect bonding

INTERVENTIONS:
Device: Quantitative Light-Induced Fluorescence — White spot lesion on the tooth surfaces detected with Quantitative Light-Induced Fluorescence Orthodontic Bonding.
Procedure: Direct bonding — The patients in the direct bonding group received a bonding procedure with a conventional composite adhesive.
  Arms: Direct Bonding; Quantitative Light-Induced Fluorescence
Procedure: Indirect bonding — For the patients in the indirect bonding group, bonding was performed with a flowable composite adhesive.
  Arms: Indirect bonding; Quantitative Light-Induced Fluorescence

SUMMARY:
The aim of this 2-arm parallel trial was to evaluate enamel demineralization after an indirect bonding technique in comparison to a direct bonding technique group using the quantitative light-induced fluorescence method. Thirty-six patients who needed fixed orthodontic treatment were randomly separated into either the direct bonding group or the indirect bonding group. Eligibility criteria included moderate crowding in the maxillary and mandibular dental arch, good oral hygiene, absence of craniofacial anomalies, no previous orthodontic treatment and no deciduous, congenitally missing or extracted teeth. Randomization was made at the start of the study with a statistical analysis program (SAS Institute Inc., Cary, NC, USA.). For the patients in the indirect bonding group, bonding was performed with a flowable composite adhesive, while the patients in the direct bonding group received a bonding procedure with a conventional composite adhesive. Records were taken using quantitative light-induced fluorescence (QLF) with a Digital Biluminator (Inspektor Research Systems, Amsterdam, the Netherlands) in the pretreatment and posttreatment examination phases. The presence and extent of lesions on the buccal surfaces of all teeth, except the molar teeth, were assessed. The fluorescence loss, lesion area and percentage of fluorescence loss were determined using the system's software. The primary outcome of this study was evaluation of the effects of bonding techniques on white spot lesion formation by using the QLF method. Random sequence generation was performed with a computerized random 1:1 allocation using block sizes of 4. It was not possible for the clinicians and their interventions to be blocked. The patients and the specialists were blinded to the treatment groups when their treatment groups were aware.

DETAILED DESCRIPTION:
This study was single center, one-blinded, 2-arm parallel, randomized clinical trial with a 1:1 allocation ratio. No changes were made to the protocol after trial commencement. Initially, 60 patients who had been referred to a tertiary clinic in Kayseri, Turkey for orthodontic treatment between October 2011 and June 2013 were assessed for eligibility by the clinicians (A.Y.). The inclusion criteria for the experiment groups in this study were mild to moderate crowding in the maxillary and mandibular dental arch, good oral hygiene, absence of craniofacial anomalies, no previous orthodontic treatment and no deciduous, congenitally missing or extracted teeth. 60 patients were examined in the trial. Thirty-six patients were divided into groups with equal numbers of patients in each group. The study was completed with 31 patients. An analysis was performed on the 15 patients in the indirect bonding group and the 16 patients in the direct bonding group. Approval for the study was obtained from the Local Ethics Committee of the Faculty of Medicine at Erciyes University in Kayseri, Turkey (11-3585). Informed consent was obtained from all the patients included in the study. The consent was obtained from those over 18 years of age directly, and from the parents of those under 18 years of age. Standard treatment records, which are photographs, dental models and radiographs, were taken in the beginning of treatment and at the end of treatment from all patients included in the study. The patients were randomly allocated to 1 of 2 treatment groups: indirect bonding and direct bonding. In the direct bonding group, after the plaque structure on the teeth was cleaned with pumice and white elastic bur were etched with 37% phosphoric acid gel (3M-Dental Products, St Paul, Minnesota, USA) for 30 seconds, the teeth were rinsed and dried with oil-free compressed air for 15 seconds. After drying the enamel surface, the liquid primer Transbond XT (3M-Unitek, Monrovia, California, USA) was applied with a small brush and spread with oil-free compressed air. Pre-adjusted metal brackets which had values for the Roth prescription were then bonded using the conventional adhesive with a standard protocol and polymerized for 3 seconds per bracket with a multiwave light-emitting diode curing light.

In the indirect bonding group, alginate was utilized to take impressions of the maxillary and mandibular arches, and hard dental stone was used to cast the dental models. Following the trimming and drying of the dental models dried, guidelines were drawn for vertical and horizontal bracket-positioning using a black pencil. The separating agent Al Cote (Dentsply Trubyte, York, Pennsylvania, USA) was administered onto the surfaces of the teeth surfaces using a brush, and the casts were left to dry. The same brackets used in the direct bonding technique were used. The composite adhesive was administered onto the base of the bracket, and the bracket was then placed onto the marked area on the tooth surface. The excess resin was carefully removed with a hand instrument. After positioning the bracket, the composite adhesive was polymerized with a multiwave light-emitting diode curing light. After positioning of the bracket on the transfer models, the composite adhesive was polymerized for 3 seconds, and a 2-layer transfer tray was prepared using translucent soft silicone and thermoformed rigid Essix Plus plastic. The base of the brackets in the transfer tray was sandblasted to remove the separating agent. A flowable composite adhesive was applied to the bracket bases, and the transfer tray was then seated on the arch segment. The composite adhesive was polymerized for 3 seconds before and after removing the transfer tray. Excessive composite adhesive remnants were then removed using a tungsten carbide bur in an air rotor instrument. For all of the patients included in the study, orthodontic treatment and recommendations for how to use toothpaste containing fluoride, how to brush their teeth and diet habits were also added to reduce the number of white spot lesions and provide better treatment. The QLF images of all patients who underwent direct and indirect bonding were taken by the same observer in the beginning of fixed orthodontic treatment (T0) and immediately after removal of the appliances (T1) at the end of the treatment period using a QLF-D Biluminator 2-camera system (Inspektor Research Systems, Amsterdam, The Netherlands).

ELIGIBILITY:
Inclusion Criteria:

* medical healthy subjects
* mild to moderate crowding in the maxillary and mandibular dental arch,
* good oral hygiene,
* absence of craniofacial anomalies,
* no previous orthodontic treatment and
* no deciduous, congenitally missing or extracted teeth.

Exclusion Criteria:

* severe crowding,
* bad oral hygiene,
* presence of craniofacial anomalies,
* previous orthodontic, orthognathic or prosthetic treatment
* presence of congenital teeth deficiency, deciduous or extracted teeth

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2011-07-28 (Actual); Primary Completion 2013-11-27 (Actual); Study Completion 2016-01-05 (Actual)

PRIMARY OUTCOMES:
White spot lesion incidence | up to 2 year
  In the indirect bonding technique group, less amount of white spot lesions are expected than the direct bonding technique in end of the treatment.

SECONDARY OUTCOMES:
Quantitative white spot lesion amounts | up to 2 year
  The QLF method gives a quantitative result, it may be used efficiently for imaging of white spot lesion formation during or after orthodontic treatment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogaard B. Prevalence of white spot lesions in 19-year-olds: a study on untreated and orthodontically treated persons 5 years after treatment. Am J Orthod Dentofacial Orthop. 1989 Nov;96(5):423-7. doi: 10.1016/0889-5406(89)90327-2. PMID 2816842
- [Background] van der Veen MH, de Josselin de Jong E. Application of quantitative light-induced fluorescence for assessing early caries lesions. Monogr Oral Sci. 2000;17:144-62. doi: 10.1159/000061639. PMID 10949838
- [Background] Sondhi A. Efficient and effective indirect bonding. Am J Orthod Dentofacial Orthop. 1999 Apr;115(4):352-9. doi: 10.1016/s0889-5406(99)70252-0. PMID 10194277
- [Result] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Result] Baysal A, Ulusoy SN, Uysal T. Evaluation of enamel demineralization in adolescents after rapid maxillary expansion using the quantitative light-induced fluorescence method: A single-center, randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2016 Nov;150(5):731-739. doi: 10.1016/j.ajodo.2016.06.014. PMID 27871699
- [Result] Yagci A, Korkmaz YN, Buyuk SK, Yagci F, Atilla AO. White spot lesion formation after treatment with full-coverage rapid maxillary expanders. Am J Orthod Dentofacial Orthop. 2016 Mar;149(3):331-8. doi: 10.1016/j.ajodo.2015.08.015. PMID 26926020
- [Result] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Derived] Atilla AO, Ozturk T, Eruz MM, Yagci A. A comparative assessment of orthodontic treatment outcomes using the quantitative light-induced fluorescence (QLF) method between direct bonding and indirect bonding techniques in adolescents: a single-centre, single-blind randomized controlled trial. Eur J Orthod. 2020 Sep 11;42(4):441-453. doi: 10.1093/ejo/cjz058. PMID 31375814